CLINICAL TRIAL: NCT02408627
Title: EEG@HOME (Phase 3a of the Project, Comparison of EEG-recordings)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Collaborators: Pilipili NV (Industry); Imec (Industry)
Responsible Party: Principal Investigator, Neurologie, Prof. dr. Kristl Vonck, University Hospital, Ghent
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Diagnostic
Other Study IDs: EC/2014/1283
Record Dates: First submitted 2015-03-31; First posted 2015-04-03 (Estimated); Last update posted 2017-11-28 (Actual); Status verified 2017-11

CONDITIONS: Epilepsy
MeSH Terms: conditions — Epilepsy | interventions — Electroencephalography

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- conventional EEG-registration type 1 (Active Comparator): conventional EEG-registration with wet bridge electrodes and conductive gel
  Interventions: Device: EEG
- conventional EEG-registration type 2 (Active Comparator): conventional EEG-registration with wet cup electrodes and collodion
  Interventions: Device: EEG
- EEG-registration with dry electrodes (Experimental): EEG-registration with dry electrodes
  Interventions: Device: EEG

INTERVENTIONS:
Device: EEG

SUMMARY:
The goal of this project is the development of an EEG-cap (min. 21 electrodes) with user-friendly active dry electrodes that meets the expectations of the users regarding comfort and esthetics, without losing sight of the functional and technical demands for recording high quality EEG signals. The purpose is to use the EEG-cap to investigate clinical neurological disorders (e.g. epilepsy). The EEG-cap could also be used at home so that hospital admission in the EMU can be avoided for some patients and an increasing number of patients can be examined.

Phase 3 of the Project will be divided into a Phase 3a and Phase 3b.

Phase 3a of the project will comprise of an EEG-registration with the different types of electrodes in epilepsy patients with prominent interictal epileptiform discharges (IEDs) on EEG. For each epilepsy patient the EEG-recording with dry electrodes will be compared to the EEG-recordings with conventionally used wet electrodes (bridge and cup electrodes). Each EEG-recording will take approximately 10 minutes.

Minimum 2 - maximum 10 epilepsy patients will be included.

There will be an visual and clinical evaluation of the EEG-signals (blinded) and a technical evaluation of the EEG-signals. User experience will also be collected.

ELIGIBILITY:
Inclusion Criteria:

* Epilepsy patients with prominent interictal epileptiform discharges (IEDs) on EEG

Exclusion Criteria:

* Epilepsy patients with no prominent interictal epileptiform discharges (IEDs) on EEG

Ages: 6 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2015-01; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
EEG signal quality (visual and clinical) (scale) | 10 minutes
EEG signal quality (technical) (signal to noise ratio) | 10 minutes
User experience (questionnaire) | 10 minutes

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Ghent, Ghent, Belgium